CLINICAL TRIAL: NCT07015333
Title: Case Review of Patients With Betel Nut-induced Oral Cancer Treated With Pembrolizumab and Cetuximab
Status: Completed | Type: Observational
Sponsor: Commonwealth Healthcare Corporation (Other)
Responsible Party: Principal Investigator, Peter Brett, MD, Director, Medical Oncology, Commonwealth Healthcare Corporation
Other Study IDs: 5-2025 Oral Cancer
Record Dates: First submitted 2025-05-25; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: pembrolizumab and cetuximab — Treatment of betel nut-induced oral cancer with pembrolizumab and cetuximab

SUMMARY:
Chart review of records of patients treated for betel nut-induced oral cancer with pembrolizumab and cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Advanced betel nut-induced oral cancer

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced betel nut-induced oral cancer
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date first treatment received until 3 months later
  Assessed by clinical measurement of largest tumor size

CONTACTS AND LOCATIONS:
Locations (1):
- CHCC, Saipan, MP, Northern Mariana Islands